CLINICAL TRIAL: NCT01049373
Title: Efficacy and Safety of Lymphdiaral Basistropfen (a Fixed Homoeopathic Remedy [HDC]) in the Treatment of Chronic Low-back Pain Considering Constitution and Diathesism: a Double Blind, Randomised, Placebo Controlled, Single-centre Study
Brief Title: Efficacy and Safety of Lymphdiaral Basistropfen (HDC) in the Treatment of Chronic Low-back Pain
Acronym: 144
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC144/03; ISRCTN88642122 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-06

CONDITIONS: Low Back Pain
Keywords: low-back; pain; chronic; constitution; diathesism; homoeopathy; fixed combination; herbal preparation; chronic low back pain lasting more than 6 months
MeSH Terms: conditions — Low Back Pain; Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lymphdiaral Basistropfen (HDC) (Experimental): HDC (Calendula mother tincture, Condurango 2X, Phytolacca 2X, Carduus marianus 1X, Chelidonium 2X, Hydrastis mother tincture, Leptandra mother tincture, Taraxacum mother tincture, Echinacea mother tincture, Lycopodium 2X, Sanguinaria mother tincture and Arsenicum album 8X), each 10 drops t.i.d. for 15 weeks.
  Interventions: Drug: HDC
- Placebo Solution (Placebo Comparator): 10 drops t.i.d. for 15 weeks
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: HDC — (Calendula mother tincture, Condurango 2X, Phytolacca 2X, Carduus marianus 1X, Chelidonium 2X, Hydrastis mother tincture, Leptandra mother tincture, Taraxacum mother tincture, Echinacea mother tincture, Lycopodium 2X, Sanguinaria mother tincture and Arsenicum album 8X),10 drops t.i.d. for 15 weeks.
  Other Names: Lymphdiaral Basistropfen
  Arms: Lymphdiaral Basistropfen (HDC)
Drug: Placebo solution — 10 drops, t.i.d, 15 weeks
  Arms: Placebo Solution

SUMMARY:
To evaluate superiority of HDC in comparison to placebo in the treatment of chronic low-back pain in relation to pain, functional impairment, quality of life, and state of health during a 15-week treatment period.

DETAILED DESCRIPTION:
Low-back pain is often provoked by inflammatory edema in the region of the facet joints. In naturopathy, a fixed homeopathic drug combination (HDC) is established in the treatment of edema and swellings. For the first time, the efficacy of HDC was investigated in the treatment of low-back pain.

Objective: To examine the efficacy and safety of HDC medication vs. placebo in the treatment of chronic low back pain considering constitution and diathesism in a double-blind, randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Aged 18 - 75 years
* Chronic low-back pain lasting at least for 6 months
* Hanover functional ability questionnaire (FFbH-R) score less than 70%
* At least one of the following diagnoses:

  1. Chronic lumbar ischialgia with or without radicular radiation
  2. Chronic degenerative lumbar syndrome
  3. Spondylarthrosis
  4. Chronic facet syndrome
  5. Lumbago with protrusion of the intervertebral disc
  6. Lumbar radiculopathy
  7. Lumbar and other intervertebral disc impairments with radiculopathy
  8. Back pain at different locations of the spine
* Written, informed consent

Exclusion Criteria:

* Participation in another clinical trial/GCP-trial within 30 days prior to screening
* Participation in this trial in an earlier time
* Treatment with lymphdiaral basistropfen within 3 month prior to enrolment
* Pregnancy and lactation
* Non-compliance
* Incapability to understand the sense of the study
* Abuse of analgesics, opiates or other drugs
* Chronic pain that are as strong as or even stronger than the pain caused by the low-back and that need to be treated with analgesics
* Malign diseases
* Pathological neurological states
* Epilepsy
* Operation of the spine within 3 month prior to enrolment
* Fractures of the spine
* Bechterew's disease
* Alcohol abuse
* Consuming diseases
* Cachexia
* Palsy of the legs or anal sphincter due to acute impairment of the intervertebral disc
* Catheterisation or CT-controlled intra-articular injection in the lumbar region
* Hypersensitivity against one of the ingredients or excipients of the study drugs or against composite plants in general
* Systemic, progressive diseases like tuberculosis, leucosis, collagenosis, multiple sclerosis, acquired immune deficiency syndrome (AIDS), human immunodeficiency virus (HIV) infection, or other auto-immune diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2003-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre M Beer, MD, PhD, Principal Investigator — Department of True Naturopathy, Blankenstein Hospital; Im Vogelsang 5-11; D-45527 Hattingen; Germany;; Juergen Kraemer, Prof, Study Director — St. Josef Hospital. Gudrunstr. 56, 44791 Bochum, Germany; Anja Braschoss, MD, Study Chair — Pascoe Pharmazeutische Praeparate GmbH
Locations (1):
- Department of Naturopathy, Blankenstein Hospital, Hattingen, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: hospital, 5.12.2003 - 5.5.2007 (first patient in / last patient out)
Pre-assignment Details: screening visit (up to one week before baseline)
Period: Overall Study
Arm/Group | Lymphdiaral Basistropfen (HDC) | Placebo Solution
Started | 112 | 109
Completed | 73 | 65
Not Completed | 39 | 44
Not completed — Protocol Violation | 9 | 9
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 9 | 4
Not completed — no evaluable study values | 9 | 21
Not completed — Other | 1 | 1
Not completed — Non-cooperation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lymphdiaral Basistropfen (HDC) | Placebo Solution | Total
Number analyzed (Participants) | 112 | 109 | 221
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 78 | 163
  >=65 years | 27 | 31 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 97 | 193
  Male | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in FFbH-R Between Screening and Week 15
Description: Hannover Functional Questionnaire (FFbH-R) As used in this study test FFbH-R is a special version of the FFbH "for close to everyday diagnostics of functional impairment by back pain". It is a patient questionnaire, which consists of 12 questions for the acquisition of functional limitations consists in activities of daily living.
  Change in FFbH-R between screening and week 15 Scale ranges from 0 (=worst) to 100(=best)
Time Frame: between screening and 15 weeks treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lymphdiaral Basistropfen (HDC) | Placebo Solution
Number analyzed (Participants) | 103 | 89
units on a scale | 8.8 (15.0) | 4.1 (15.3)
Statistical Analysis 1: Comparison: Lymphdiaral Basistropfen (HDC) vs Placebo Solution; Test type: Superiority or Other; p = 0.0426, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in FFbH-R Between Screening and 2 Weeks
Description: Hannover Functional Questionnaire (FFbH-R) As used in this study test FFbH-R is a special version of the FFbH "for close to everyday diagnostics of functional impairment by back pain". It is a patient questionnaire, which consists of 12 questions for the acquisition of functional limitations consists in activities of daily living.
  Change in FFbH-R between screening and 2 weeks Scale ranges from 0 (=worst) to 100(=best)
Time Frame: between screening and 2 weeks treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lymphdiaral Basistropfen (HDC) | Placebo Solution
Number analyzed (Participants) | 103 | 89
units on a scale | 3.9 (12.8) | 0.6 (12.7)
Statistical Analysis 1: Comparison: Lymphdiaral Basistropfen (HDC) vs Placebo Solution; Test type: Superiority or Other; p = 0.0757, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Pain Score (SES), Subscale "Sensoric Pain"
Description: Pain Perception Scale (SES) The SES is a patient questionnaire, which consists of 24 questions, both the affective (14 questions) and sensoric (10 questions) depict aspects.
  Difference between V1 minus V-1 in the subscale "sensoric pain" Scale ranges from 10(=best) to 40(=worst)
Time Frame: following 2 weeks treatment
Population: Only patients with assessable values at present time point were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- LYMPHDIARAL (HDC): HDC (Calendula mother tincture, Condurango 2X, Phytolacca 2X, Carduus marianus 1X, Chelidonium 2X, Hydrastis mother tincture, Leptandra mother tincture, Taraxacum mother tincture, Echinacea mother tincture, Lycopodium 2X, Sanguinaria mother tincture and Arsenicum album 8X), each 10 drops t.i.d. for 15 weeks.
Arm/Group | LYMPHDIARAL (HDC) | Placebo Solution
Number analyzed (Participants) | 99 | 86
units on a scale | -4.2 (7.5) | -1.8 (5.4)
Statistical Analysis 1: Comparison: LYMPHDIARAL (HDC) vs Placebo Solution; Test type: Superiority or Other; p = 0.0465, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Pain Score (SES), Subscale "Sensoric Pain"
Description: Pain Perception Scale (SES) The SES is a patient questionnaire, which consists of 24 questions, both the affective (14 questions) and sensoric (10 questions) depict aspects.
  Difference between screening and 15 weeks in the subscale "sensoric pain" Scale ranges from 10(=best) to 40(=worst)
Time Frame: following 15 weeks treatment
Population: Only patients with assessable values at present time point were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LYMPHDIARAL (HDC) | PLACEBO Solution
Number analyzed (Participants) | 70 | 62
units on a scale | -5.4 (6.8) | -3.9 (7.3)
Statistical Analysis 1: Comparison: LYMPHDIARAL (HDC) vs PLACEBO Solution; Test type: Superiority or Other; p = 0.04443, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Strength of Pain (Visual Analog Scale VAS)
Time Frame: following 2 weeks treatment
Reporting Status: Not Posted

6. Secondary Outcome: Change in Strength of Pain (Visual Analog Scale VAS)
Time Frame: following 15 weeks treatment
Reporting Status: Not Posted

7. Secondary Outcome: Change in State of Health (BF-S)
Time Frame: following 2 weeks treatment
Reporting Status: Not Posted

8. Secondary Outcome: Change in State of Health (BF-S)
Time Frame: following 15 weeks treatment
Reporting Status: Not Posted

9. Secondary Outcome: Change in Oswestry Score
Time Frame: following 2 weeks treatment
Reporting Status: Not Posted

10. Secondary Outcome: Change in Oswestry Score
Time Frame: following 15 weeks treatment
Reporting Status: Not Posted

11. Secondary Outcome: Change in Short Form Health Survey 12 Items (SF-12)
Time Frame: following 2 weeks treatment
Reporting Status: Not Posted

12. Secondary Outcome: Change in Short Form Health Survey 12 Items (SF-12) Ment
Time Frame: following 15 weeks treat
Reporting Status: Not Posted

13. Secondary Outcome: Correlation of Efficacy With the Constitutional Type of the Patient, Measured by the Hattinger Constitutional Manual (HKM) and the Hattinger Constitutional Questionnaire (HKF)
Time Frame: following 15 weeks treatment
Reporting Status: Not Posted

14. Secondary Outcome: Amount of Analgesics Used
Time Frame: 15 weeks treatment
Reporting Status: Not Posted

15. Secondary Outcome: Number of Days With Incapability to Work
Time Frame: 15 weeks treatment
Reporting Status: Not Posted

16. Secondary Outcome: Number of ADRs
Description: frequency of ADR with a probable or possible causal relationship
Time Frame: within 15 weeks treatment
Measure: Number; unit: adverse reactions
Arm/Group | LYMPHDIARAL (HDC) | Placebo Solution
Number analyzed (Participants) | 112 | 109
adverse reactions | 8 | 7

ADVERSE EVENTS:
Time Frame: from 2003-Dec-05 to 2007-May-05
Arm/Group | Lymphdiaral Basistropfen (HDC) | Placebo Solution
Serious Adverse Events (participants affected / at risk) | 6/112 | 7/109
Other Adverse Events (participants affected / at risk) | 43/112 | 39/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphdiaral Basistropfen (HDC) (N=112) | Placebo Solution (N=109)
Athroscopy (Investigations) | 1 (1) | 0 (0) — unlikely
Depression (Psychiatric disorders) | 1 (1) | 0 (0) — not related
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — not related
Mental disoerder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0) — not related
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) — not related
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — possible
Musculosskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — not related
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — not related
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1) — not related
Intestinal operation (Surgical and medical procedures) | 0 (0) | 1 (1) — not related
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) — not related
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphdiaral Basistropfen (HDC) (N=112) | Placebo Solution (N=109)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 2 (2)
Dizziness (Nervous system disorders) | 5 (5) | 9 (9)
Erythema (Skin and subcutaneous tissue disorders) | 5 (7) | 2 (2)
Headache (Nervous system disorders) | 21 (25) | 18 (21)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (11) | 6 (8)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less